CLINICAL TRIAL: NCT06977776
Title: Evaluation of the Effectiveness of a Web-Based Osteoporosis Awareness Training Program Based on the Health Belief Model in Female University Students With Osteoporosis Risk
Brief Title: Effectiveness of a Web-Based Osteoporosis Awareness Education Program Based on the Health Belief Model Among Female University Students at Risk
Acronym: Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Meryem Gürler, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05.10.2023- 326/07
Record Dates: First submitted 2025-04-22; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Osteoporosis; Women; Young Individuals; Risk Factors
Keywords: Osteoporosis; Health Belief Model (HBM); Female university students; Awareness
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: Intervention Group: The group that will receive Osteoporosis Awareness Training.
  Control Group: The group receiving no intervention. The intervention group will receive Osteoporosis Awareness Training. The control group will be given pre-test and post-test without training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Group Receiving Osteoporosis Awareness Education
  Interventions: Behavioral: Web-Based Osteoporosis Awareness Training Based on Health Belief Model
- Control Group (No Intervention): Only pre-test and post-test will be applied.

INTERVENTIONS:
Behavioral: Web-Based Osteoporosis Awareness Training Based on Health Belief Model — This study presents a web-based osteoporosis awareness training based on the health belief model. The training is designed to provide information about the risks of osteoporosis, ways of prevention and healthy lifestyle habits. Participants will be taught about the importance of calcium intake, the benefits of exercise and osteoporosis prevention methods. The training process will be supported by interactive content and individual counseling sessions offered through the website and participants will be provided with the opportunity to consolidate their knowledge.
  Arms: Intervention Group

SUMMARY:
Study Title: Evaluation of the Effectiveness of a Web-Based Osteoporosis Awareness Training Program Based on the Health Belief Model in Female University Students with Osteoporosis Risk

Background: Osteoporosis is a common disease worldwide, leading to a high risk of fractures, especially in women. According to World Health Organization (WHO) criteria, osteoporosis is defined as a bone mineral density (BMD) of 2.5 standard deviations or less in young, healthy women. Osteoporosis usually progresses asymptomatically and interferes with activities of daily living, leading to high mortality and morbidity rates. Furthermore, the cost of osteoporosis is estimated at 12.2-17.9 billion dollars per year worldwide. Therefore, raising awareness and adopting a healthy lifestyle are important to reduce the risk of osteoporosis among young women.

Objective: This study aims to evaluate the effectiveness of a web-based educational program based on the health belief model for female university students at risk for osteoporosis.

Method: The study will be conducted with a randomized controlled design. Participants will be enrolled in a web-based training program aiming to increase their knowledge about osteoporosis risk factors, preventive health behaviors and healthy lifestyle. The effectiveness of the training program will be evaluated in terms of participants' level of knowledge about osteoporosis, health beliefs and behavioral changes.

Target Population: Female university students aged 18-24 years, who are at risk of osteoporosis.

Expected Outcomes: The training program is expected to result in a positive change in participants' osteoporosis knowledge, health beliefs and preventive behaviors. Furthermore, it is important to disseminate such trainings among young women as an effective strategy for osteoporosis prevention.

Conclusion: This study will constitute an important step towards osteoporosis prevention by aiming to increase young women's knowledge about osteoporosis, strengthen their health beliefs and improve their healthy living habits. Proving the effectiveness of the training program will shed light on the development and implementation of similar health education programs in the future.

Keywords: Osteoporosis, Health Belief Model, Education Program, Female University Students, Awareness, Preventive Health Behaviors.

DETAILED DESCRIPTION:
Osteoporosis is a common disease worldwide. According to the World Health Organization criteria, osteoporosis is defined as a bone mineral density (BMD) 2.5 standard deviations or more below the mean value (T score < - 2.5 SD) for young, healthy women. It is known as a silent disease leading to millions of osteoporotic fractures annually worldwide. The World Health Organization (WHO) has declared osteoporosis as the main enemy of human health, along with heart attack, stroke and cancer.

Osteoporosis can progress without symptoms for a long time. It is also known as a problem with high mortality, morbidity and cost as well as preventing the individual's daily life activities. Symptoms of osteoporosis include deterioration of body posture, back and lower back pain and fractures. Fractures can be caused by minor traumas and are most common in the spine, wrist and hip bones.

Risk factors for osteoporosis are divided into modifiable and non-modifiable causes. Modifiable risk factors include dietary calcium deficiency, physical inactivity, low body mass index, smoking and alcohol consumption and long-term medication use. Gender, age, race, fair skin and genetic characteristics are considered as non-modifiable osteoporosis risk factors. Although osteoporosis is a problem for both genders, most of the research on osteoporosis focuses on women. This is because women are more likely to develop osteoporosis and subsequent fractures than men. This is because men develop more bone mass during growth and more muscle mass that provides skeletal integration. In addition, men do not go through menopause and have a shorter life expectancy than women. Therefore, they have less time to develop the disease.

In a meta-analysis conducted in five continents, the prevalence of osteoporosis was reported to be 18.3% worldwide (prevalence of osteoporosis in women worldwide is 23.1% and prevalence of osteoporosis in men worldwide is 11.7%). In 2018, another systematic review and meta-analysis based on World Health Organization (WHO) diagnostic criteria in the Eastern Mediterranean showed that the prevalence of osteoporosis was 24.4% between 2000 and 2017 (prevalence of osteoporosis was 24.4% in women and 20.5% in men). Fracture is the most important complication of osteoporosis. In the United States, the lifetime probability of osteoporosis-related fracture for every woman and every man is estimated to be one in two and one in five, respectively. Among European women, the lifetime probability of hip fracture is reported to be 7-25% and major osteoporotic fractures at age 50 are reported to be approximately 50%. In Turkey, osteopenia was found in half and osteoporosis in ¼ of people over the age of 50, and the rate of osteoporosis-related hip fractures has increased over the years. In Turkey, hip fractures are more common in urban areas and in physically inactive people (TOD). In addition, a study reported that 6.9% of Turkish women aged 18-49 years have a moderate to high risk of osteoporosis. The direct medical cost of osteoporosis is estimated to be 12.2-17.9 billion dollars per year worldwide.

In women, physical inactivity, reduced calcium and vitamin D intake, age, menstrual cycle changes, smoking and alcohol consumption impair bone mass density, which is shaped early in life, doubles by age 20 and shrinks rapidly by age 50. Therefore, it is important for young women to maintain bone mass early in life (in the first three decades of life), increase women's knowledge about the disease and adopt a healthy lifestyle to reduce the risk of osteoporosis among women.

Osteoporosis knowledge and awareness has been an important topic in different international studies. Most of these studies have found a lack of knowledge and awareness about osteoporosis in women of different age groups, as well as lack of exercise and calcium intake practices and less self-efficacy or confidence in preventive behaviors. Most of these studies focused on knowledge and found that there is insufficient knowledge about osteoporosis, especially among female university students, and that although they have positive self-efficacy towards exercise and negative self-efficacy towards calcium intake, their knowledge and perceptions are not shown in their behaviors. This age group, which coincides with the university period, is important. Because bone density doubles at the age of 20. Many university students may not have reached peak bone mass. Behaviors developed with sufficient knowledge can bring the bone mass to the level it will reach. Therefore, increasing awareness and knowledge about osteoporosis is thought to be of great value in improving bone health in this age group.

Osteoporosis is a disease that can be prevented by raising awareness of the society since childhood. For this purpose, children and young people should gain proper nutrition and exercise behaviors, which are social strategies to prevent osteoporosis. In developing health behaviors for osteoporosis, not only information but also health beliefs of individuals are important. In preventing osteoporosis, the health belief model is effective in education to increase individuals' perceptions of osteoporosis health, perceptions of benefits and motivation and to decrease their perceptions of barriers. This model directs individuals to engage in desired health behaviors as a motivational tool. Therefore, it is used to protect and improve the health of young women at risk of osteoporosis.

ELIGIBILITY:
Inclusion Criteria:-Be a woman

* To be a first year undergraduate student,
* To be studying outside the field of health,
* Not being an international student,
* Not to have graduated from a high school related to health,
* No previous education on osteoporosis,
* Not having problems with musculoskeletal system, cardiopulmonary system and other systems that would prevent exercise,
* Being in the medium and high risk group according to the osteporosis risk assessment,

Exclusion Criteria: -Wanting to leave the research at any stage of the research,

* Not fully participating in the Osteoporosis Awareness Training program,
* Participants who incompletely completed the data collection forms will be excluded from the study.

Ages: 18 Weeks to 25 Weeks | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — female
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Osteoporosis Knowledge Test (OBT) Score | Pre-training (day 0) and post-training (after 8 weeks and after 12 weeks)
  A scale used to assess the level of knowledge participants have about osteoporosis. Scores before and after the training will be compared.

SECONDARY OUTCOMES:
Osteoporosis Health Belief Scale (OHBS) Score | Pre-training (day 0) and post-training (after 8 weeks and 12 weeks).
  A scale used to measure participants' health beliefs about osteoporosis. Scores before and after the training will be compared.
Osteoporosis Self-Efficacy-Efficacy Scale (OSESES) Score | Pre-training (day 0) and post-training (after 8 weeks and 12 weeks).
  A scale used to assess participants' perception of self-efficacy related to osteoporosis. Scores before and after the training will be compared.
Results of the Calcium-Specific Food Frequency Survey (CFSF) | Pre-training (day 0) and post-training (after 8 weeks and 12 weeks).
  A questionnaire used to assess the frequency of calcium intake of the participants. It will be compared before and after the training.
International Physical Activity Questionnaire (IPAQ) Results | Pre-training (day 0) and post-training (after 8 weeks and 12 weeks).
  A questionnaire used to assess the physical activity level of the participants. It will be compared before and after the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi evran Üniversitesi, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is aimed to share the results and data of the study with other researchers to contribute to the literature on osteoporosis awareness and the effectiveness of education programs. The shared data will pave the way for more comprehensive studies on osteoporosis prevention and health education. It will also enable studies to be conducted that will increase the effectiveness of the health belief model and test its applicability in different demographic groups. Sharing data will help to develop new strategies aimed at increasing awareness of osteoporosis by promoting scientific collaboration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code